CLINICAL TRIAL: NCT05210114
Title: Cutaneous Hydration Assessment in Sickle Cell Disease
Brief Title: Cutaneous Hydration Assessment in SCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Enrico Novelli (Other)
Responsible Party: Sponsor-Investigator, Enrico Novelli, Associate Professor and Section Chief - Classical Hematology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY21090014
Record Dates: First submitted 2021-12-26; First posted 2022-01-27 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Skin Hydration Sensor (Experimental)
  Interventions: Device: Skin Hydration Sensor

INTERVENTIONS:
Device: Skin Hydration Sensor — The device is a skin hydration sensor. The sensor is placed on the skin at the inner arm. It is non-invasive and measures in seconds the percent water content of the dermis by quantifying its dielectric constant.
  Other Names: Delfin MoistureMeterEpiD

SUMMARY:
This study will validate the diagnostic accuracy of a cutaneous hydration sensor. This sensor will also be evaluated for its feasibility as a point-of-care device for the assessment of hydration status and its potential to guide hydration therapy in patients with sickle cell disease (SCD).

DETAILED DESCRIPTION:
Vaso-occlusive episodes (VOE) are the leading cause of hospitalization for patients with SCD. Intravenous fluid replacement is one of the cornerstones of management of VOE in the emergency department and throughout hospitalization. However, there are no evidence-based guidelines specifying the optimal administration of maintenance fluids. Overly aggressive hydration therapy imparts the risk of hypervolemia and pulmonary edema, which may lead to acute chest syndrome and death. Thus, a reliable biomarker is needed to gauge hydration status and guide fluid replacement strategies with the goal of achieving euvolemia.

The investigators propose a point-of-care test that may inform management (e.g., bolus vs. continuous infusion of maintenance intravenous fluid), and prevent over- or under-hydration. For this purpose, investigators seek to validate the diagnostic accuracy of a cutaneous hydration sensor, Delfin MoistureMeterEpiD (a non-significant risk device) and evaluate its feasibility as a point-of-care device for the assessment of hydration status and potentially guide hydration therapy in patients with SCD. Investigators will measure skin hydration in the clinic when participants are at baseline state of health. Skin hydration before and after fluid resuscitation therapy in patients with vaso-occlusive crisis (VOC) or VOE will also be assessed. Blood and urine will be collected to compare assessments of skin hydration with laboratory biomarkers of hypertonicity and red blood cell dehydration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Sickle Cell Disease (genotypes SS, SC, Sß-thalassemia, SD, SOArab)
* Participants must be ≥12-years old
* Participants that provide legally effective consent to all study procedures

Exclusion Criteria:

* Participants under 12-years old
* Participants being treated with experimental therapies in clinical trials

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dermal water content measurements in SCD participants at baseline state of health | During a regularly scheduled clinic appointment, approximately 2 hours
  Delfin MoistureMeterEpiD hydration sensor will be used to measure dermal water content in 20 participants at 1 time point.
Dermal water content measurements before fluid resuscitation in SCD participants with VOC or VOE | During a VOC or VOE event before IV fluid resuscitation, approximately 2 hours
  Delfin MoistureMeterEpiD hydration sensor will be used to measure dermal water content in 10 participants.
Dermal water content measurements after fluid resuscitation in SCD participants with VOC or VOE | During a VOC or VOE event after IV fluid resuscitation, approximately 2 hours
  Delfin MoistureMeterEpiD hydration sensor will be used to measure dermal water content in 10 participants.
Clinical dehydration assessments in SCD participants | At a regularly scheduled clinical appointment, approximately 2 hours
  Clinical assessment of dehydration will be ascertained by administering the 10-point Clinical Dehydration Scale (CDS). CDS uses clinical characteristics (general appearance, eyes, mucous membranes, and tears), each of which are scored 0, 1, or 2 for a total score of 0 to 8, with 0 representing no dehydration; 1 to 4, some dehydration; and 5 to 8, moderate/severe dehydration. It will be administered at 1 time point in 20 participants.
Measurement of serum osmolality as a laboratory biomarker of dehydration in SCD participants | At a regularly scheduled clinical appointment, approximately 2 hours
  Serum osmolality values of >290 milliosmol/kg is considered abnormal. It will be measured at 1 timepoint in 20 participants.
Measurement of hyperadhesion as a laboratory biomarker of dehydration in SCD participants | At a regularly scheduled clinical appointment, approximately 2 hours
  As a marker of hyperadhesion capillary transit time will be measured using capillary mimicking microfluidic channels. It will be measured at 1 timepoint in 20 participants.
Measurement of elongation index as a cellular biomarker of dehydration in SCD participants | At a regularly scheduled clinical appointment, approximately 2 hours
  Cellular dehydration marker, the elongation index, will be measured by ektacytometry. It will be measured at 1 timepoint in 20 participants.
Measurement of point of sickling as a biomarker of dehydration in SCD participants | At a regularly scheduled clinical appointment, approximately 2 hours
  Point of sickling, a cellular dehydration biomarker, will be measured by ektacytometry. It will be measured at 1 timepoint in 20 participants.
Measurement of urine osmolality as a laboratory biomarker of dehydration in SCD participants | At a regularly scheduled clinical appointment, approximately 2 hours
  Urine osmolality values <450 milliosmol/kg is considered abnormal in adults without fluid restrictions. It will be measured at 1 timepoint in 20 participants.
Measurement of serum osmolality as a laboratory biomarker of dehydration before resuscitation therapy in SCD participants with VOC or VOE | During a VOC or VOE event before resuscitation therapy, approximately 2 hours
  Serum osmolality values of >290 milliosmol/kg is considered abnormal. It will be measured at 1 timepoint in 10 participants.
Measurement of serum osmolality as a laboratory biomarker of dehydration after fluid resuscitation therapy in SCD participants with VOC or VOE | During a VOC or VOE event after fluid resuscitation therapy, approximately 2 hours
  Serum osmolality values of >290 milliosmol/kg is considered abnormal. It will be measured at 1 timepoint in 10 participants.
Measurement of hyperadhesion as a laboratory biomarker of dehydration before fluid resuscitation therapy in SCD participants with VOC or VOE | During a VOC or VOE event before fluid resuscitation therapy, approximately 2 hours
  As a marker of hyperadhesion, capillary transit time will be measured using capillary mimicking microfluidic channels. It will be measured at 1 timepoint in 10 participants.
Measurement of hyperadhesion as a laboratory biomarker of dehydration after fluid resuscitation therapy in SCD participants with VOC or VOE | During a VOC or VOE event after fluid resuscitation therapy, approximately 2 hours
  As a marker of hyperadhesion, capillary transit time will be measured using capillary mimicking microfluidic channels. It will be measured at 1 timepoint in 10 participants.
Measurement of elongation index as a cellular biomarker of dehydration before resuscitation therapy in SCD participants with VOC or VOE | During a VOC or VOE event before fluid resuscitation, approximately 2 hours
  Cellular dehydration marker, the elongation index, will be measured by ektacytometry. It will be measured at 1 timepoint in 10 participants.
Measurement of elongation index as a cellular biomarker of dehydration after fluid resuscitation therapy in SCD participants with VOC or VOE | During a VOC or VOE event after fluid resuscitation therapy, approximately 2 hours
  Cellular dehydration marker, the elongation index will be measured by ektacytometry. It will be measured at 1 timepoint in 10 participants.
Measurement of point of sickling as a cellular biomarker of dehydration before fluid resuscitation therapy in SCD participants with VOC or VOE | During a VOC or VOE event before fluid resuscitation therapy, approximately 2 hours
  Cellular dehydration marker, the elongation index will be measured by ektacytometry. It will be measured at 1 timepoint in 10 participants.
Measurement of point of sickling as a cellular biomarker of dehydration after fluid resuscitation therapy in SCD participants with VOC or VOE | During a VOC or VOE event after fluid resuscitation therapy, approximately 2 hours
  Cellular dehydration marker, the elongation index will be measured by ektacytometry. It will be measured at 1 timepoint in 10 participants.
Measurement of urine osmolality as laboratory biomarkers of dehydration before fluid resuscitation therapy in SCD participants with VOC or VOE | During a VOC or VOE event before fluid resuscitation therapy, approximately 2 hours
  Urine osmolality values <450 milliosmol/kg is considered abnormal in adults without fluid restrictions. It will be measured at 1 timepoint in 10 participants.
Measurement of urine osmolality as laboratory biomarkers of dehydration after fluid resuscitation therapy in SCD participants with VOC or VOE | During a VOC or VOE event after fluid resuscitation therapy, approximately 2 hours
  Urine osmolality values <450 milliosmol/kg is considered abnormal in adults without fluid restrictions. It will be measured at 1 timepoint in 10 participants.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Novelli, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Sickle Cell Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No